CLINICAL TRIAL: NCT04702490
Title: A Phase 2A Study to Evaluate MET409 Alone or in Combination With Empagliflozin in Patients With Type 2 Diabetes Mellitus (T2DM) and Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study to Evaluate MET409 Alone or in Combination With Empagliflozin in Patients With Type 2 Diabetes and NASH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Metacrine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET409-201
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: NASH; NASH - Nonalcoholic Steatohepatitis; Type 2 Diabetes; Diabetes Type 2; Diabetes; Fatty Liver; Fatty Liver, Nonalcoholic; NAFLD
Keywords: NASH; FXR; Fatty Liver; Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus; Fatty Liver | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MET409 A (Experimental): MET409 Active (50mg)
  Interventions: Drug: MET409 Active
- MET409 P (Placebo Comparator): MET409 Placebo (50mg)
  Interventions: Drug: MET409 Placebo
- MET409A +Open-Label Empagliflozin (Experimental): MET409 Active (50mg) + Empagliflozin (10mg)
  Interventions: Drug: MET409 Active; Drug: Empagliflozin
- MET409P +Open-Label Empagliflozin (Placebo Comparator): MET409 Placebo (50mg) + Empagliflozin (10mg)
  Interventions: Drug: MET409 Placebo; Drug: Empagliflozin

INTERVENTIONS:
Drug: MET409 Active — MET409 Active (50mg)
  Arms: MET409 A; MET409A +Open-Label Empagliflozin
Drug: MET409 Placebo — MET409 Placebo (50mg)
  Arms: MET409 P; MET409P +Open-Label Empagliflozin
Drug: Empagliflozin — Empagliflozin (10mg)
  Arms: MET409A +Open-Label Empagliflozin; MET409P +Open-Label Empagliflozin

SUMMARY:
A randomized, multi-center study evaluating MET409 (50 mg) alone or in combination with empagliflozin (10 mg) for 12 weeks. Assignment to MET409 will be double-blind and placebo-controlled. Empagliflozin will be incorporated into two of the treatment arms in an open-label manner.

DETAILED DESCRIPTION:
Subjects assigned to receive empagliflozin will be dosed at 10 mg per day for the duration of the study.

Approximately 30 subjects will be enrolled per treatment arm.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females 18 through 75 years of age.
* Diagnosis of NASH based on NAFLD Activity Score (NAS) ≥ 4 with at least 1 point in each of steatosis, inflammation, and ballooning; Magnetic Resonance Elastography (MRE) showing kPa ≥ 2.61 or a multiparametric MRI (ie, LiverMultiScan) showing iron-corrected T1(cT1) > 830 ms within 6 months of enrollment; or Transient elastography (TE, FibroScan) with liver stiffness ≥ 8.5 kPa and controlled attenuation parameter (CAP) > 300 dB/m obtained within 3 months of enrollment.
* Liver fat content ≥ 8% measured by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) during screening.
* Diagnosis of T2DM for ≤ 10 years, with hemoglobin A1c ≤ 10.0% during screening, stable and controlled with diet or treatment for at least 3 months.

Key Exclusion Criteria:

* History of significant liver disease (eg, alcoholic liver disease, viral hepatitis, etc.) or liver transplant.
* Presence of cirrhosis on any prior liver biopsy (stage 4 fibrosis).
* Excessive consumption of alcohol.
* Use of any insulin (injectable or inhaled), SGLT-2 inhibitor or glucagon-like peptide 1 (GLP-1, injectable or oral) products for > 7 days within 3 months of screening.
* Weight loss > 10% in the 6 months prior to screening or > 5% during screening.
* Use of drugs historically associated with causing NAFLD for more than 4 consecutive weeks within 12 months prior to screening.
* Concomitant use of drugs that are strong or moderate CYP3A4 inhibitors.
* Concomitant consumption of grapefruit juice with the study drug.
* History of diabetic ketoacidosis (DKA) within 1 month prior to the Screening Visit, or more than 2 episodes within 6 months prior to the Screening Visit.
* History of > 2 episodes of urosepsis or pyelonephritis within 5 years of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of MET409 with or without empagliflozin (incidence of adverse events) | Up to 28 days after last dose
  Incidence of Treatment-emergent adverse events, incidence of clinically significant changes in vital signs, abnormal laboratory safety tests, and abnormal ECGs.

SECONDARY OUTCOMES:
Pharmacological activity of MET409 alone or in combination with empagliflozin | 16 weeks
  Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF)
Pharmacokinetic profile of MET409 alone or in combination with empagliflozin | 12 weeks
  Cmax
Pharmacokinetic profile of MET409 alone or in combination with empagliflozin | 12 weeks
  tmax
Pharmacokinetic profile of MET409 alone or in combination with empagliflozin | 12 weeks
  AUClast
Pharmacodynamic profile of MET409 alone or in combination with empagliflozin | 16 weeks
  Bile acid precursor : C4 (7αhydroxy-4-cholesten-3-one)
Pharmacodynamic profile of MET409 alone or in combination with empagliflozin | 16 weeks
  Bile acid precursor : Fibroblast growth factor 19 (FGF19)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert C Chen, MD, Study Chair — Metacrine, Inc.
Locations (2):
- United States (2):
  - Metacrine Investigative Site, Fort Myers, Florida
  - Metacrine Investigative Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Metacrine — https://www.metacrine.com/